CLINICAL TRIAL: NCT01027949
Title: An Open-Label Extension Trial of UT-15C SR in Subjects With Pulmonary Arterial Hypertension
Brief Title: An Open-Label Extension Trial of UT-15C Sustained-release (SR) in Subjects With Pulmonary Arterial Hypertension
Acronym: FREEDOM-EXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-304
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

ARMS (1):
- Oral Treprostinil (Experimental): Subjects from previous studies TDE-PH-202 (NCT01104870), TDE-PH-203 (NCT01477333), and TDE-PH-205 (NCT01588405), TDE-PH-301 (NCT00325442), TDE-PH-302 (NCT00325403), or TDE PH-308 (NCT00887978). Subjects were instructed to take the appropriate amount of 0.125, 0.25, 0.5, 1, and/or 2.5 mg tablets based upon their prescribed dose. Investigators were instructed to increase the dose of oral treprostinil in the absence of dose limiting drug-related AEs to ensure each subject received the optimal clinical dose throughout the study
  Interventions: Drug: Oral Treprostinil

INTERVENTIONS:
Drug: Oral Treprostinil — Oral sustained release tablet, twice or thrice daily. Open label study with active drug, no other intervention arms.
  Other Names: Treprostinil diethanolamine, treprostinil diolamine; UT-15C

SUMMARY:
This study provided/continued to provide oral treprostinil (UT-15C SR; treprostinil diethanolamine) to eligible subjects who participated in Studies TDE-PH-202, TDE-PH-203, TDE-PH-205, TDE-PH-301, TDE-PH-302, and TDE-PH-308. The study assessed the long term safety of oral treprostinil and the effect of continued treatment with oral treprostinil on exercise capacity after 1 year of treatment.

DETAILED DESCRIPTION:
This was an international, multicenter, open-label study designed to provide oral treprostinil for eligible subjects who participated in Studies TDE-PH-301, TDE-PH-302, TDE-PH-308, TDE-PH-202, TDE PH 203, and TDE-PH-205. Subjects randomly allocated to receive oral treprostinil in Studies TDE-PH-301, TDE-PH-302, or TDE-PH-308 and enrolled in this open-label study completed visits at Months 6, 12, 24, 36, and yearly visits thereafter. Subjects randomly allocated to receive placebo in Studies TDE-PH-301, TDE-PH-302, or TDE-PH-308 completed visits at Months 3, 6, 12, 24, 36, and yearly visits thereafter. Subjects that transitioned from Studies TDE-PH-202, TDE-PH-203, and TDE-PH-205 (that had an open-label study design) followed the regimen for subjects receiving oral treprostinil. A 6-Minute Walk Test (6MWT) and Borg dyspnea score were conducted at the visit which occurred 12 months after the subject's first exposure to oral treprostinil.

Adverse events (AEs) were reported continuously throughout the study; any AEs ongoing at the time of discharge from Studies TDE PH-301, TDE PH-302, TDE-PH-308, TDE-PH-202, TDE-PH-203, and TDE-PH-205 were recorded as AEs and marked as "ongoing from previous study" in the subject's electronic Case Report Form (eCRF). Study drug dosing and pulmonary arterial hypertension (PAH) concomitant medication usage were assessed at each scheduled study visit and recorded in the subject's eCRF.

ELIGIBILITY:
Inclusion Criteria:

1. The subject remained on study drug and completed all assessments during the Treatment Phase of the previous study (TDE-PH-202, TDE-PH-203, TDE-PH-205, TDE-PH-301, TDE PH-302, or TDE-PH-308) OR the subject permanently discontinued study drug during the Treatment Phase of the previous study due to clinical worsening (as defined in the protocol of the previous study), completed premature termination assessments prior to discontinuing study drug, completed all remaining scheduled study visits, AND received placebo during the Treatment Phase of the previous studies OR the subject was randomized into Group 1 or Group 2 in Study TDE PH 202, permanently discontinued study drug during the 12-week Treatment Phase due to clinical worsening, completed all premature termination assessments prior to discontinuing study drug, and completed all remaining scheduled study visits and assessments (with the exception of the hemodynamic measurements) through Week 12. Such subjects should have started treatment with oral treprostinil in the open-label study at 0.25 mg twice daily (BID).
2. The subject voluntarily gave informed consent to participate in the study.
3. Women of childbearing potential includes any female who had experienced menarche and who had not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or was not postmenopausal (defined as amenorrhea for at least 12 consecutive months). Sexually active women of childbearing potential must have used 2 effective forms of contraception during the length of the study. Medically acceptable forms of effective contraception included: (1) approved hormonal contraceptives (such as birth control pills), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, (3) an intrauterine device, (4) partner vasectomy, or (5) abstinence. Males participating in the study must have used a condom during the length of the study, and for at least 48 hours after discontinuing study medication. Protocol Amendment A.1AU included the required assessment for Austrian subjects to perform urine pregnancy tests every 4 weeks during the study.

Exclusion Criteria:

1. The subject permanently discontinued study drug during the previous study (TDE PH 202, TDE-PH-203, TDE PH 205, TDE-PH-301, TDE-PH-302, or TDE PH 308) due to treatment-related adverse events (AEs).
2. The subject permanently discontinued study drug during the Treatment Phase of the previous study (TDE-PH-202, TDE-PH-203, TDE-PH-205, TDE-PH-301, TDE-PH-302, or TDE-PH-308) due to clinical worsening (as defined in those study protocols) and did not undergo premature termination assessments prior to discontinuing study drug, and/or did not complete all remaining study visits through the final scheduled visit.
3. The subject prematurely discontinued study drug during the Treatment Phase of the previous study due to clinical worsening (as defined in those study protocols), completed premature termination assessments prior to discontinuing study drug, completed all remaining scheduled study visits AND received oral treprostinil during the Treatment Phase of the previous study (TDE PH-202, TDE-PH-203, TDE-PH-301, TDE-PH-302, or TDE PH-308). Subjects enrolled in Study TDE-PH-202 who were randomized into the individual maximum tolerated dose (iMTD) group who clinically worsened could not participate. Subjects who permanently discontinued study drug during the 12-week Treatment Phase due to treatment-related AEs were not eligible even if they completed all remaining scheduled study visits. Subjects who permanently discontinued study drug during the 12 week Treatment Phase and did not undergo premature termination assessments prior to discontinuing study drug and/or who did not complete all remaining study visits through the Week 12 visit were also not eligible.
4. The subject developed any concurrent illness or condition during the conduct of the previous study, including but not restricted to: sleep apnea, chronic renal insufficiency, anemia, uncontrolled systemic hypertension, or left sided heart disease, unless their physician felt that entry into this study would not be detrimental to their overall health.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 894 (Actual)
Dates: Start 2007-01-16 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (135):
- United States (61):
  - The Kirklin Clinic, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University Medical Center, Tucson, Arizona
  - University of Arizona Clinical and Translational Science (CATS) Research Center, Tucson, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford University, Pulmonary and Critical Care Medicine, Stanford, California
  - Harbor-UCLA Medical Center, Torrance, California
  - The Children's Hospital, Aurora, Colorado
  - University of Colorado Health Science Center, Aurora, Colorado
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - The Emory Clinic, Atlanta, Georgia
  - The University of Chicago Hospitals, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - Mary Parkes Center, Rochester, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Carl and Ethyl Linder Center for Research and Education at the Christ Church, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - Legacy Pulmonary Clinic, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Medical School, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Australia (4):
  - The Prince Charles Hospital, Chermside West
  - Heart/Lung Transplant Unit - St. Vincent's Hospital, Darlinghurst
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
- Austria (3):
  - Medizininische Universitaet Wien, Vienna
  - Universitaetsklinik für Innere Medizin Innsbruck, Vienna
  - Medical University Graz, Wein
- Belgium (2):
  - Department of Cardiology Erasme University Hospital, Brussels
  - University Hospital Gasthuisberg, Leuven
- Canada (6):
  - Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Coastal Health Authority Vancouver General Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - London Health Sciences Center Victoria Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- China (3):
  - Beijing Shijitan Hospital, Cadres Respiratory Department, Beijing
  - Peking Union Medical College Hospital, Respiratory Medicine Department, Beijing
  - Shanghai Pulmonary Hospital, Respiratory Medicine Department, Shanghai
- France (8):
  - Service Chirurgie Thoracique, Hôpital Haut Levêque, Pessac, Pessac Cedex
  - PMAC, Clinique de Pneumologie, Bernin
  - Centre d'Investigation Clinique Hôpital La Cavale Blanche - CHU Brest, Brest
  - Hospital Antoine Beclere, Clamart
  - Hospital Claude Huriez, Lille
  - Hôpital Louis Pradel, Lyon
  - CHU Arnaud de Villeneuve - Service maladies respiratoires, Montpellier
  - Service de Pneumologie Centre de Competence pour l'HTAP- Pole des Voies Respiratoires Hôpital Larrey, Toulouse
- Germany (8):
  - Universitätsklinikum Dresden Abtl. Pneumologie, Dresden
  - University Hospital Greifswald, Greifswald
  - DRK Kliniken Berlin Köpenick, Hamburg
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinkium Köln Klinik III für Innere Medizin, Hamburg
  - Zentrum für Lungenhochdruck Thoraxklinik am Universitätsklinikum Heidelberg, Hamburg
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Dept. of Internal Medicine III University Heidelberg, Heidelberg
- India (11):
  - Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - Narayana Hrudayalaya Hospitals, Bangalore, Karnataka
  - Asian Heart Institute & Research Centre Pvt. Ltd., Mumbai, Maharashtra
  - Poona Hospital and Research Centre, Pune, Maharashtra
  - Life Care Institute of Medical Sciences & Research, Ahmedabad
  - Sri Ramachandra Medical College & Research Institute, Chennai
  - G. Kuppuswamy Naidu Memorial Hospital, Coimbatore
  - PRIME Hospitals, Hyderabad
  - Sir Ganga Ram Hospital, New Delhi
  - Ruby Hall Clinic, Pune
  - Queen's NRI Hospital, Visakhapatnam
- Pulmonary Hypertension Unit Centre for Lung Health Mater Misericordiae University Hospital, Dublin, Ireland
- Israel (5):
  - Rambam Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Pulmonary Institute Rabin Medical Center (Belinson Kampus), Petah Tikva
  - Pulmonary Institute Chaim Sheba Medical Center, Ramat Gan
- Italy (4):
  - Policlinico S. Orsola Malpighi - Università degli studi di Bologna, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale Monaldi - Cotugno-CTO Cardiologia S.U.N., Naples
  - Azienda Ospedaliera di Rilievo Nazionale Monaldi - Cotugno-CTO Cardiologia S.U.N., Napoli
  - Dipartimento di Scienze Cardiovascolari, Respiratorie e Morfologiche, Rome
- Mexico (3):
  - Instituto Nacional de Cardiologia, Mexico City
  - Hospital Universitario de la UANL, Monterrey
  - Unidad de Investigacion Clinica en Medicina S.C., Monterrey
- Netherlands (2):
  - Radboud University Nijmegen Medical Center, Amsterdam
  - VU Medish Centrum, Amsterdam
- Poland (3):
  - Klinika Chorób Serca i Naczyń, Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Europejskie Centrum Zdrowia Otwock, Warsaw
  - Oddzial Kardiologiczny, Wroclaw
- Servico de Cardiologia Hospital de Santa Marta, Lisbon, Portugal
- Auxilio Mutuo Hospital CardioPulmonary Research Center, Guaynabo, Puerto Rico
- Spain (3):
  - Hospital Clínic I Provincial, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
- Skane University Hospital, Lund, Sweden
- United Kingdom (5):
  - Papworth Hospital, Cambridge
  - Papworth Hospital NHS Foundation Trust, Glasgow
  - Royal Free Hospital, London
  - Freeman Hospital, Newcastle
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Baseline values for demographic parameters were defined and collected in the same manner for subjects who received either placebo or oral treprostinil in the preceding studies. Note that Studies TDE-PH-202 (NCT01104870), TDE-PH-203 (NCT01477333), and TDE-PH-205 (NCT01588405) had an open-label design; therefore, all Baseline demographic parameters were based on values collected at the time of enrollment in the previous study.
Pre-assignment Details: Subjects eligible for TDE-PH-304 previously participated in Studies TDE-PH-202 (NCT01104870), TDE-PH-203 (NCT01477333), and TDE-PH-205 (NCT01588405), TDE-PH-301 (NCT00325442), TDE-PH-302 (NCT00325403), or TDE PH-308 (NCT00887978).
Groups:
- Oral Treprostinil: Subjects eligible for TDE-PH-304 previously participated in Studies TDE-PH-202 (NCT01104870), TDE-PH-203 (NCT01477333), and TDE-PH-205 (NCT01588405), TDE-PH-301 (NCT00325442), TDE-PH-302 (NCT00325403), or TDE PH-308 (NCT00887978)
Period: Overall Study
Arm/Group | Oral Treprostinil
Started | 894
Completed | 208
Not Completed | 686
Not completed — Death | 174
Not completed — Progressive Disease | 163
Not completed — Adverse Event | 172
Not completed — Withdrawal by Subject | 113
Not completed — Lost to Follow-up | 17
Not completed — Protocol Violation | 13
Not completed — PI Decision | 8
Not completed — Limited Study Drug Effectiveness | 7
Not completed — Non-compliance with Study Procedures | 7
Not completed — Lung Transplant | 5
Not completed — Unable to Tolerate Study Drug | 2
Not completed — Use of Excluded Medication | 2
Not completed — Patient Self-discontinuation | 1
Not completed — Pregnancy | 1
Not completed — Surgery | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the study.
Groups:
- Oral Treprostinil: Subjects eligible for TDE-PH-304 previously participated in Studies TDE PH-202, TDE-PH-203, TDE-PH-205, TDE-PH-301, TDE-PH-302, or TDE PH-308.
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 894
Age, Continuous [Mean (Full Range); unit: years] | 47.7 [12 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 696
  Male | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83
  Not Hispanic or Latino | 809
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 34
  Asian | 219
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 46
  White | 589
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 1
  United States | 436
  United Kingdom | 27
  Portugal | 1
  India | 79
  Spain | 6
  Canada | 19
  Austria | 7
  Netherlands | 15
  Sweden | 2
  Belgium | 6
  Ireland | 2
  Poland | 16
  Italy | 13
  Mexico | 38
  Israel | 22
  Australia | 44
  France | 22
  Germany | 14
  China | 124
PAH Etiology [Count of Participants; unit: Participants]
  Idiopathic Pulmonary Arterial Hypertension/ Heritable Pulmonary Arterial Hypertension | 608
  Collagen Vascular Disease | 224
  Other | 60
  Missing | 2
World Health Organization (WHO) Functional Class [Count of Participants; unit: Participants] — WHO PAH Groups are defined as follows. The groups are categorical classifications for subjects with PAH and are not a severity grading system.
  I = Pulmonary Arterial Hypertension II = Pulmonary Hypertension due to left heart disease III = Pulmonary Hypertension due to lung disease IV = Pulmonary Hypertension due to blood clots in the lungs V = Blood and other rare disorders that lead to Pulmonary Hypertension
  Participants
    I | 18
    II | 298
    III | 527
    IV | 11
    Missing | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Capacity at Month 12
Description: Assess the effect of continued therapy with oral treprostinil on exercise capacity as assessed by the change from Baseline in 6-Minute Walk Test (6MWT) after 1 year of treatment. The 6MWT is the clinical standard for assessing subject functional status in the treatment of PAH and has been considered an objective measure of subject functional status by the American Thoracic Society. The distance a subject can walk in 6 minutes is recorded in meters.
Time Frame: From First Visit (Visit 1) to Month 12
Population: All subjects enrolled in the study with Baseline and matched follow-up 6MWTs.
Measure: Median (Full Range); unit: meters
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 572
meters | 22.0 [-345.0 to 282.0]

ADVERSE EVENTS:
Time Frame: From the time of subject enrollment until exit from the study (up to 13 years).
Arm/Group | Oral Treprostinil
All-Cause Mortality (participants affected / at risk) | 174/894
Serious Adverse Events (participants affected / at risk) | 547/894
Other Adverse Events (participants affected / at risk) | 890/894
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil (N=894)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 129 (147)
Right ventricular failure (Cardiac disorders) | 129 (188)
Pneumonia (Infections and infestations) | 63 (76)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (51)
Acute kidney injury (Renal and urinary disorders) | 37 (48)
Cardiac failure (Cardiac disorders) | 36 (43)
Syncope (Nervous system disorders) | 30 (33)
Anaemia (Blood and lymphatic system disorders) | 28 (32)
Chest pain (General disorders) | 28 (33)
Hypotension (Vascular disorders) | 23 (26)
Fluid overload (Metabolism and nutrition disorders) | 21 (27)
Cardiac failure congestive (Cardiac disorders) | 19 (26)
Atrial fibrillation (Cardiac disorders) | 15 (18)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Sudden death (General disorders) | 15 (15)
Atrial flutter (Cardiac disorders) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 13 (15)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (13)
Bronchitis (Infections and infestations) | 11 (13)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 (17)
Lower respiratory tract infection (Infections and infestations) | 11 (12)
Nausea (Gastrointestinal disorders) | 11 (11)
Gastritis (Gastrointestinal disorders) | 10 (11)
Gastroenteritis (Gastrointestinal disorders) | 10 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Sepsis (Infections and infestations) | 10 (11)
Vomiting (Gastrointestinal disorders) | 10 (10)
Sudden cardiac death (General disorders) | 10 (10)
Cardiogenic shock (Cardiac disorders) | 9 (10)
Dehydration (Metabolism and nutrition disorders) | 9 (13)
Supraventricular tachycardia (Cardiac disorders) | 9 (13)
Ascites (Gastrointestinal disorders) | 8 (9)
Cellulitis (Infections and infestations) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 8 (8)
Cardiac arrest (Cardiac disorders) | 7 (7)
Death (General disorders) | 7 (7)
Headache (Nervous system disorders) | 7 (7)
Urinary tract infection (Infections and infestations) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Abortion induced (Surgical and medical procedures) | 6 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 (6)
Pericardial effusion (Cardiac disorders) | 6 (7)
Pyrexia (General disorders) | 6 (6)
Renal failure (Renal and urinary disorders) | 6 (7)
Subdural haematoma (Injury, poisoning and procedural complications) | 6 (6)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6)
Deep vein thrombosis (Vascular disorders) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5)
Oedema peripheral (General disorders) | 5 (6)
Palpitations (Cardiac disorders) | 5 (5)
Pancytopenia (Blood and lymphatic system disorders) | 5 (5)
Presyncope (Nervous system disorders) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Mental status changes (Psychiatric disorders) | 5 (5)
Non-cardiac chest pain (General disorders) | 5 (6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Fluid retention (Metabolism and nutrition disorders) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 (5)
Ventricular extrasystoles (Cardiac disorders) | 4 (4)
Large intestine polyp (Gastrointestinal disorders) | 4 (4)
Disease progression (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory tract infection (Infections and infestations) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Asthenia (General disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Generalised oedema (General disorders) | 3 (4)
Haematuria (Renal and urinary disorders) | 3 (5)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
International normalised ratio increased (Investigations) | 3 (3)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Melaena (Gastrointestinal disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Portal hypertension (Hepatobiliary disorders) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Viral infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 3 (3)
Hepatic enzyme increased (Investigations) | 3 (4)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 3 (3)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Appendicitis (Infections and infestations) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2)
Blood glucose decreased (Investigations) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Chest discomfort (General disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cor pulmonale (Cardiac disorders) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Flushing (Vascular disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2)
Hypopituitarism (Endocrine disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lupus nephritis (Renal and urinary disorders) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Osteomyelitis (Infections and infestations) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (3)
Rectal ulcer (Gastrointestinal disorders) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Shock (Vascular disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3)
Suicidal ideation (Psychiatric disorders) | 2 (4)
Tachycardia (Cardiac disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2)
Typhoid fever (Infections and infestations) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Visual impairment (Eye disorders) | 2 (2)
General physical health deterioration (General disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure high output (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Carotid body tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Coma hepatic (Nervous system disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cyanosis central (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (6)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypersplenism (Blood and lymphatic system disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Impaired healing (General disorders) | 1 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
International normalised ratio abnormal (Investigations) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Mass (General disorders) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
Ovarian rupture (Reproductive system and breast disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small cell lung cancer limited stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1)
Evans syndrome (Blood and lymphatic system disorders) | 1 (1)
Sepsis syndrome (Infections and infestations) | 1 (1)
Central line infection (Infections and infestations) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1)
Palliative care (Surgical and medical procedures) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Angiodysplasia (Vascular disorders) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paracentesis (Investigations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1)
Balloon atrial septostomy (Surgical and medical procedures) | 1 (1)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Pseudomonas bronchitis (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1)
Vascular compression (Vascular disorders) | 1 (1)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil (N=894)
Flushing (Vascular disorders) | 416 (499)
Hypotension (Vascular disorders) | 79 (91)
Fatigue (General disorders) | 201 (228)
Oedema peripheral (General disorders) | 192 (240)
Chest pain (General disorders) | 135 (180)
Pain (General disorders) | 97 (102)
Pyrexia (General disorders) | 83 (100)
Chest discomfort (General disorders) | 57 (70)
Asthenia (General disorders) | 51 (64)
Oedema (General disorders) | 43 (44)
Insomnia (Psychiatric disorders) | 95 (98)
Anxiety (Psychiatric disorders) | 57 (60)
Depression (Psychiatric disorders) | 56 (59)
Weight decreased (Investigations) | 47 (49)
Dizziness (Cardiac disorders) | 248 (320)
Palpitations (Cardiac disorders) | 145 (175)
Right ventricular failure (Cardiac disorders) | 136 (202)
Cardiac failure (Cardiac disorders) | 42 (54)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 207 (294)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 190 (215)
Cough (Respiratory, thoracic and mediastinal disorders) | 159 (202)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 98 (103)
Epistais (Respiratory, thoracic and mediastinal disorders) | 77 (88)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 45 (57)
Anaemia (Blood and lymphatic system disorders) | 84 (112)
Headache (Nervous system disorders) | 698 (994)
Syncope (Nervous system disorders) | 101 (141)
Presyncope (Nervous system disorders) | 51 (55)
Diarrhoea (Gastrointestinal disorders) | 592 (808)
Nausea (Gastrointestinal disorders) | 505 (673)
Vomiting (Gastrointestinal disorders) | 349 (485)
Abdominal pain (Gastrointestinal disorders) | 121 (144)
Abdominal pain upper (Gastrointestinal disorders) | 97 (111)
Abdominal distension (Gastrointestinal disorders) | 92 (102)
Dyspepsia (Gastrointestinal disorders) | 92 (95)
Constipation (Gastrointestinal disorders) | 65 (74)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 46 (48)
Abdominal discomfort (Gastrointestinal disorders) | 45 (48)
Acute kidney injury (Renal and urinary disorders) | 52 (69)
Rash (Skin and subcutaneous tissue disorders) | 79 (87)
Pruritus (Skin and subcutaneous tissue disorders) | 43 (50)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 313 (360)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 255 (337)
Arthralgia (Musculoskeletal and connective tissue disorders) | 140 (163)
Myalgia (Musculoskeletal and connective tissue disorders) | 123 (143)
Back pain (Musculoskeletal and connective tissue disorders) | 105 (127)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 64 (71)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 42 (44)
Decreased appetite (Metabolism and nutrition disorders) | 129 (142)
Hypokalaemia (Metabolism and nutrition disorders) | 94 (119)
Fluid overload (Metabolism and nutrition disorders) | 44 (58)
Fluid retention (Metabolism and nutrition disorders) | 43 (54)
Upper respiratory tract infection (Infections and infestations) | 222 (334)
Nasopharyngitis (Infections and infestations) | 185 (316)
Bronchitis (Infections and infestations) | 103 (153)
Pneumonia (Infections and infestations) | 94 (118)
Urinary tract infection (Infections and infestations) | 89 (115)
Sinusitis (Infections and infestations) | 80 (108)
Influenza (Infections and infestations) | 54 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2013-03-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT01027949/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT01027949/SAP_001.pdf